CLINICAL TRIAL: NCT02280811
Title: A Phase I/II Study of T Cell Receptor Gene Therapy Targeting HPV-16 E6 for HPV-Associated Cancers
Brief Title: T Cell Receptor Immunotherapy Targeting HPV-16 E6 for HPV-Associated Cancers
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Christian S. Hinrichs, M.D., Principal Investigator, National Institutes of Health Clinical Center (CC)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 150005; 15-C-0005
Record Dates: First submitted 2014-10-30; First posted 2014-11-03 (Estimated); Results first posted 2017-08-02 (Actual); Last update posted 2017-09-06 (Actual); Status verified 2017-08

CONDITIONS: Vaginal Cancer; Cervical Cancer; Anal Cancer; Penile Cancer; Oropharyngeal Cancer
Keywords: HPV positive; Metastatic; Diet; Screening; Risk Factors; Colorectal adenoma; Refractory; Immunotherapy; Reproductive Cancers
MeSH Terms: conditions — Vaginal Neoplasms; Uterine Cervical Neoplasms; Anus Neoplasms; Penile Neoplasms; Oropharyngeal Neoplasms; Neoplasm Metastasis | interventions — fludarabine; fludarabine phosphate; Cyclophosphamide; aldesleukin; Interleukin-2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- T Cell Receptor Immunotherapy (Experimental): patients will receive cyclophosphamide and fludarabine followed by infusion of the human papilloma virus (HPV) E6 T cell receptor (TCR), followed by high dose aldesleukin
  Interventions: Drug: Fludarabine; Drug: Cyclophosphamide; Biological: E6 TCR; Drug: Aldesleukin

INTERVENTIONS:
Drug: Fludarabine — Patients will receive Fludarabine 25 mg/m^2/day for 5 days.
  Other Names: Fludara
Drug: Cyclophosphamide — Patients will receive Cyclophosphamide 60 mg/kg/day x 2 days
  Other Names: Cytoxan
Biological: E6 TCR — On day 0, cells will be infused intravenously (IV) over 20-30 minute (between 1 and 4 days after the last dose of fludarabine)
Drug: Aldesleukin — Aldesleukin 720,000 IU/kg IV (based on total body weight) over 15 minutes approximately every 8 hours beginning within 24 hours of cell infusion and continuing for up to 5 days (maximum of 15 doses).
  Other Names: IL-2

SUMMARY:
Background:

The National Cancer Institute (NCI) Surgery Branch has developed an experimental therapy for treating patients with cancer that involves taking white blood cells from the patient, growing them in the laboratory in large numbers, genetically modifying these specific cells with a type of virus (retrovirus) to attack only the tumor cells, and then giving the cells back to the patient. This type of therapy is called gene transfer. Researchers want to test this on human papilloma virus (HPV)-associated cancers.

Objective:

- The purpose of this study is to determine a safe number of these cells to infuse and to see if these particular tumor-fighting cells (Anti-HPV E6) can shrink tumors associated with HPV and test the toxicity of this treatment.

Eligibility:

- Adults age 18-66 with an HPV-16-associated cancer.

Design:

* Work up stage: Patients will be seen as an outpatient at the National Institutes of Health (NIH) clinical Center and undergo a history and physical examination, scans, x-rays, lab tests, and other tests as needed
* Leukapheresis: If the patients meet all of the requirements for the study they will undergo leukapheresis to obtain white blood cells to make the anti HPV E6 cells. {Leukapheresis is a common procedure, which removes only the white blood cells from the patient.}
* Treatment: Once their cells have grown, the patients will be admitted to the hospital for the conditioning chemotherapy, the anti HPV E6 cells and aldesleukin. They will stay in the hospital for about 4 weeks for the treatment.

Follow up: Patients will return to the clinic for a physical exam, review of side effects, lab tests, and scans about every 1-3 months for the first year, and then every 6 months to 1 year as long as their tumors are shrinking. Follow up visits take up to 2 days.

DETAILED DESCRIPTION:
BACKGROUND:

* Metastatic or refractory/recurrent human papillomavirus (HPV)-16+ cancers (cervical, vulvar, vaginal, penile, anal, and oropharyngeal cancers) are incurable and poorly palliated by standard therapies.
* HPV-16+ cancers constitutively express the HPV-16 E6 oncoprotein, which is absent from healthy human tissues.
* Administration of T cell receptor (TCR) gene engineered T cells can induce objective tumor responses in certain malignancies.
* T cells genetically engineered with a TCR targeting HPV-16 E6 (E6 TCR) display specific reactivity against human leukocyte antigen serotype within HLA-A A serotype group (HLA-A2+), HPV-16+ target cells.

OBJECTIVES:

Primary Objective

* To determine a safe dose of administration of autologous T cells transduced with an anti-HPV-16 E6 TCR and aldesleukin to patients following a nonmyeloablative but lymphodepleting preparative regimen.
* To determine the objective tumor response rate (Complete or Partial Response) and duration in patients with metastatic or recurrent/refractory HPV-16+ cancers treated with this regimen.

ELIGIBILITY:

* Patients greater than or equal to 18 years old and less than or equal to 70 years old with metastatic or refractory/recurrent HPV-16+ cancer.
* Prior first line systemic therapy is required unless the patient declines standard treatment.
* Patients must be HLA-A 02:01-positive.

DESIGN:

* Patients will receive a non-myeloablative lymphocyte-depleting preparative regimen of cyclophosphamide and fludarabine
* On day 0 patients will receive transduced lymphocytes and then begin high dose aldesleukin
* The study will begin with a phase I dose escalation. After the maximum tolerated dose (MTD) cell dose has been determined, the patients will be enrolled into the phase II portion of the study.
* Clinical and immunologic response will be evaluated about 4 to 6 weeks after treatment and then about every 1-6 months until disease progression
* Following a dose escalation phase of 9 to 18 patients, initially 21 evaluable patients will be enrolled in the phase II portion of the study. If 0 to 1 of the 21 patients experiences a clinical response, then no further patients will be enrolled. If 2 or more of the first 21 evaluable patients enrolled have a clinical response, then accrual will continue until a total of 41 evaluable patients have been enrolled. The accrual ceiling will be set at 61 patients. Provided that about 1 patient every 6 weeks will be enrolled onto this trial, approximately 4 years may be needed to accrue the maximum number of patients.

ELIGIBILITY:
-INCLUSION CRITERIA

1. Measurable metastatic or refractory/recurrent human papilloma virus (HPV-16+) cancer (determined by in situ hybridization (ISH) or a polymerase chain reaction (PCR)-based test).
2. Patients must be human leukocyte antigens (HLA-A) 02:01-positive.
3. All patients must have received prior first line standard therapy or declined standard therapy, and have been either non-responders (progressive disease) or have recurred.
4. Patients with 3 or fewer brain metastases that are less than 1 cm in diameter and asymptomatic are eligible. Lesions that have been treated with stereotactic radiosurgery must be clinically stable for 1 month after treatment for the patient to be eligible. Patients with surgically resected brain metastases are eligible.
5. Greater than or equal to 18 years of age and less than or equal to 70 years of age.
6. Able to understand and sign the Informed Consent Document.
7. Willing to sign durable power of attorney
8. Clinical performance status of Eastern Cooperative Oncology Group (ECOG) 0 or 1.
9. Life expectancy of greater than 3 months.
10. Patients of both genders must be willing to practice birth control from the time of enrollment on this study up to 4 months after treatment. Patients must be willing to undergo testing for HPV-16 prior to becoming pregnant.
11. Women of child bearing potential must have a negative pregnancy test because of the potentially dangerous effects of the treatment on the fetus.
12. Serology:

    * Seronegative for human immunodeficiency virus (HIV) antibody. (The experimental treatment being evaluated in this protocol depends on an intact immune system. Patients who are HIV seropositive can have decreased immune-competence and thus are less responsive to the experimental treatment and more susceptible to its toxicities.)
    * Seronegative for hepatitis B antigen, and seronegative for hepatitis C antibody. If hepatitis C antibody test is positive, then the patient must be tested for the presence of antigen by reverse transcription polymerase chain reaction (RT-PCR) and be hepatitis C virus ribonucleic acid (HCV RNA) negative.
13. Hematology:

    * Absolute neutrophil count greater than 1000/mm^3 without the support of filgrastim.
    * White blood cell (WBC) greater than or equal to 3000/mm^3
    * Platelet count greater than or equal 100,000/mm^3
    * Hemoglobin greater than 8.0 g/dL
14. Chemistry:

    * Serum alanine aminotransferase (ALT)/aspartate aminotransferase (AST) less than or equal to 2.5 times the upper limit of normal
    * Serum creatinine less than or equal to 1.6 mg/dL
    * Total bilirubin less than or equal to to 1.5 mg/dL, except in patients with Gilberts Syndrome who must have a total bilirubin less than 3.0 mg/dL
15. More than 4 weeks must have elapsed since any prior systemic therapy at the time the patient receives the preparative regimen.

EXCLUSION CRITERIA:

1. Women of childbearing potential who are pregnant or breastfeeding. There are potentially dangerous side effects of the treatment on the fetus or infant.
2. Active systemic infections (for e.g.: requiring anti-infective treatment), coagulation disorders or other active major medical illnesses of the cardiovascular, respiratory or immune system, as evidenced by a positive stress thallium or comparable test, myocardial infarction, cardiac arrhythmias, obstructive or restrictive pulmonary disease.
3. Any form of primary immunodeficiency (such as Severe Combined Immunodeficiency Disease).
4. Concurrent opportunistic infections (The experimental treatment being evaluated in this protocol depends on an intact immune system. Patients who have decreased immune competence may be less responsive to the experimental treatment and more susceptible to its toxicities).
5. Concurrent systemic steroid therapy.
6. History of severe immediate hypersensitivity reaction to cyclophosphamide or fludarabine.
7. History of coronary revascularization or ischemic symptoms.
8. Documented left ventricular ejection fraction (LVEF) of less than or equal to 45% tested. The following patients will undergo cardiac evaluations

a. clinically significant atrial and/or ventricular arrhythmias including but not limited to: atrial fibrillation, ventricular tachycardia, second or third degree heart block or

b. age greater than or equal 60 years old

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2014-10-14 (Actual); Primary Completion 2016-06-28 (Actual); Study Completion 2016-06-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christian S Hinrichs, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rosenberg SA. Raising the bar: the curative potential of human cancer immunotherapy. Sci Transl Med. 2012 Mar 28;4(127):127ps8. doi: 10.1126/scitranslmed.3003634. PMID 22461638
- [Background] Hinrichs CS, Rosenberg SA. Exploiting the curative potential of adoptive T-cell therapy for cancer. Immunol Rev. 2014 Jan;257(1):56-71. doi: 10.1111/imr.12132. PMID 24329789
- [Background] Chaturvedi AK, Engels EA, Pfeiffer RM, Hernandez BY, Xiao W, Kim E, Jiang B, Goodman MT, Sibug-Saber M, Cozen W, Liu L, Lynch CF, Wentzensen N, Jordan RC, Altekruse S, Anderson WF, Rosenberg PS, Gillison ML. Human papillomavirus and rising oropharyngeal cancer incidence in the United States. J Clin Oncol. 2011 Nov 10;29(32):4294-301. doi: 10.1200/JCO.2011.36.4596. Epub 2011 Oct 3. PMID 21969503
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2015-C-0005.html

RESULTS

PARTICIPANT FLOW:
Groups:
- HPV-16 E6 mTCR PBL 1x10^9 + HD IL-2; HPV-16 E6 mTCR PBL 1x10^10 + HD IL-2; HPV-16 E6 mTCR PBL 1x10^11 + HD IL-2; HPV-16 E6 mTCR PBL >1x10^11 up to 2x10^11 + HD IL-2: patients will receive cyclophosphamide and fludarabine followed by infusion of the human papilloma virus (HPV) E6 T cell receptor (TCR), followed by high dose aldesleukin
  Fludarabine: Patients will receive Fludarabine 25 mg/m^2/day for 5 days.
  Cyclophosphamide: Patients will receive Cyclophosphamide 60 mg/kg/day x 2 days
  E6 TCR: On day 0, cells will be infused intravenously (IV) over 20-30 minute (between 1 and 4 days after the last dose of fludarabine)
  Aldesleukin: Aldesleukin 720,000 IU/kg IV (based on total body weight) over 15 minutes approximately every 8 hours beginning within 24 hours of cell infusion and continuing for up to 5 days (maximum of 15 doses).
- HPV-16 E6 mTCR PBL MTD + HD IL-2: This is the phase 2 arm that was treated at the MTD determined in the phase 1 portion.
  patients will receive cyclophosphamide and fludarabine followed by infusion of the human papilloma virus (HPV) E6 T cell receptor (TCR), followed by high dose aldesleukin
  Fludarabine: Patients will receive Fludarabine 25 mg/m^2/day for 5 days.
  Cyclophosphamide: Patients will receive Cyclophosphamide 60 mg/kg/day x 2 days
  E6 TCR: On day 0, cells will be infused intravenously (IV) over 20-30 minute (between 1 and 4 days after the last dose of fludarabine)
  Aldesleukin: Aldesleukin 720,000 IU/kg IV (based on total body weight) over 15 minutes approximately every 8 hours beginning within 24 hours of cell infusion and continuing for up to 5 days (maximum of 15 doses).
Period: Drug Administration
Arm/Group | HPV-16 E6 mTCR PBL 1x10^9 + HD IL-2 | HPV-16 E6 mTCR PBL 1x10^10 + HD IL-2 | HPV-16 E6 mTCR PBL 1x10^11 + HD IL-2 | HPV-16 E6 mTCR PBL >1x10^11 up to 2x10^11 + HD IL-2 | HPV-16 E6 mTCR PBL MTD + HD IL-2
Started | 1 | 2 | 1 | 6 | 2
Completed | 1 | 2 | 1 | 6 | 2
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Retreated at the MTD
Arm/Group | HPV-16 E6 mTCR PBL 1x10^9 + HD IL-2 | HPV-16 E6 mTCR PBL 1x10^10 + HD IL-2 | HPV-16 E6 mTCR PBL 1x10^11 + HD IL-2 | HPV-16 E6 mTCR PBL >1x10^11 up to 2x10^11 + HD IL-2 | HPV-16 E6 mTCR PBL MTD + HD IL-2
Started | 0 | 0 | 0 | 0 | 1 (Patient originally started in Grp1(HPV-16 E6mTCR PBL 1x10^9+HD IL-2) and was retreated at the MTD.)
Completed | 0 | 0 | 0 | 0 | 1
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- HPV-16 E6 mTCR PBL MTD + HD IL-2: patients will receive cyclophosphamide and fludarabine followed by infusion of the human papilloma virus (HPV) E6 T cell receptor (TCR), followed by high dose aldesleukin
  Fludarabine: Patients will receive Fludarabine 25 mg/m^2/day for 5 days.
  Cyclophosphamide: Patients will receive Cyclophosphamide 60 mg/kg/day x 2 days
  E6 TCR: On day 0, cells will be infused intravenously (IV) over 20-30 minute (between 1 and 4 days after the last dose of fludarabine)
  Aldesleukin: Aldesleukin 720,000 IU/kg IV (based on total body weight) over 15 minutes approximately every 8 hours beginning within 24 hours of cell infusion and continuing for up to 5 days (maximum of 15 doses).
- Total: Total of all reporting groups
Arm/Group | HPV-16 E6 mTCR PBL 1x10^9 + HD IL-2 | HPV-16 E6 mTCR PBL 1x10^10 + HD IL-2 | HPV-16 E6 mTCR PBL 1x10^11 + HD IL-2 | HPV-16 E6 mTCR PBL >1x10^11 up to 2x10^11 + HD IL-2 | HPV-16 E6 mTCR PBL MTD + HD IL-2 | Total
Number analyzed (Participants) | 1 | 2 | 1 | 6 | 2 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 2 | 1 | 5 | 1 | 10
  >=65 years | 0 | 0 | 0 | 1 | 1 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.0 (0) | 34.5 (3.5) | 46.0 (0) | 53.5 (12.5) | 60.0 (14.1) | 50.5 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 1 | 5 | 1 | 10
  Male | 0 | 0 | 0 | 1 | 1 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 0 | 0 | 1
  Not Hispanic or Latino | 1 | 1 | 1 | 6 | 2 | 11
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0
  White | 1 | 1 | 1 | 6 | 2 | 11
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 0 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 1 | 2 | 1 | 6 | 2 | 12
Baseline Cancer Types [Count of Participants; unit: Participants]
  Cervical | 0 | 2 | 1 | 3 | 0 | 6
  Anal | 0 | 0 | 0 | 2 | 2 | 4
  Oropharyngeal | 0 | 0 | 0 | 1 | 0 | 1
  Vaginal | 1 | 0 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD)
Description: The MTD is the highest dose at which ≤1 of 6 patients experienced a dose limiting toxicity (DLT) or the highest dose level studied if DLTs are not observed at any of the dose levels.
Time Frame: participants were followed for the duration of hospital stay, an average of 3 weeks
Measure: Number; unit: # of cells x 10^11
Groups:
- All Treated Subjects: All treated subjects who received at least one dose of human papilloma virus (HPV)-16 E6 monoclonal T cell receptor (mTCR) peripheral blood lymphocytes (PBL) 1x10^9, 1x10^10,1x10^11, >1x10^11 up to 2x10^11 + high-dose (HD) interleukin 2 (IL-2) were included.
Arm/Group | All Treated Subjects
Number analyzed (Participants) | 10
# of cells x 10^11 | 2

2. Primary Outcome: Objective Tumor Response Rate (Complete or Partial Response)
Description: Objective tumor response rate is defined as the number of participants with a complete or partial response per the Response Evaluation Criteria in Solid Tumors (RECIST) v1.0. Complete response is disappearance of all target lesions. Partial response is at least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum LD.
Time Frame: 4 years
Measure: Number; unit: participants
Arm/Group | HPV-16 E6 mTCR PBL 1x10^9 + HD IL-2 | HPV-16 E6 mTCR PBL 1x10^10 + HD IL-2 | HPV-16 E6 mTCR PBL 1x10^11 + HD IL-2 | HPV-16 E6 mTCR PBL >1x10^11 up to 2x10^11 + HD IL-2 | HPV-16 E6 mTCR PBL MTD + HD IL-2
Number analyzed (Participants) | 1 | 2 | 1 | 6 | 2
participants
  Complete Response (CR) | 0 | 0 | 0 | 0 | 0
  Partial Response (PR) | 0 | 0 | 0 | 2 | 0

3. Primary Outcome: Duration of Response
Description: Duration of response is measured from the time measurement criteria are met for complete response or partial response (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented (taking as reference for progressive disease the smallest measurements recorded since the treatment started). Response is assessed by the Response Evaluation Criteria in Solid Tumors (RECIST) v1.0. Complete response is disappearance of all target lesions. Partial response is at least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum LD. Progression is at least a 20% increase in the sum of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions.
Time Frame: up to one year
Measure: Mean (95% Confidence Interval); unit: months
Arm/Group | HPV-16 E6 mTCR PBL 1x10^9 + HD IL-2 | HPV-16 E6 mTCR PBL 1x10^10 + HD IL-2 | HPV-16 E6 mTCR PBL 1x10^11 + HD IL-2 | HPV-16 E6 mTCR PBL >1x10^11 up to 2x10^11 + HD IL-2 | HPV-16 E6 mTCR PBL MTD + HD IL-2
Number analyzed (Participants) | 1 | 2 | 1 | 6 | 2
months | NA [NA to NA] — Participants had no responses. | NA [NA to NA] — Participants had no responses. | NA [NA to NA] — Participants had no responses. | 1.5 [0 to 6] | NA [NA to NA] — Participants had no responses.

4. Secondary Outcome: Number of Participants With Serious and Non-serious Adverse Events
Description: Here is the number of participants with serious and non-serious adverse events assessed by the Common Terminology Criteria in Adverse Events (CTCAE v3.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: 19 months and 7 days
Measure: Count of Participants; unit: Participants
Arm/Group | HPV-16 E6 mTCR PBL 1x10^9 + HD IL-2 | HPV-16 E6 mTCR PBL 1x10^10 + HD IL-2 | HPV-16 E6 mTCR PBL 1x10^11 + HD IL-2 | HPV-16 E6 mTCR PBL >1x10^11 up to 2x10^11 + HD IL-2 | HPV-16 E6 mTCR PBL MTD + HD IL-2
Number analyzed (Participants) | 1 | 2 | 1 | 6 | 2
Participants | 1 | 2 | 1 | 6 | 2

5. Secondary Outcome: Number of Participants With a Dose Limiting Toxicity (DLT)
Description: A dose limiting toxicity is all Grade 3 and greater toxicities with the exception of myelosuppression, defined as lymphopenia, neutropenia, decreased hemoglobin, and thrombocytopenia, due to chemotherapy preparative regimen. Aldesleukin expected toxicities as defined in Appendix 2 and 3 of the protocol. Expected chemotherapy toxicities as defined in the pharmaceutical information section. Immediate hypersensitivity reactions (excluding symptomatic bronchospasm and grade 4 hypotension) occurring within 2 hours of cell infusion (related to cell infusion) that are reversible to a grade 2 or less within 24 hours of cell administration with standard therapy. Grade 3 fever. Events that are clearly related to the patient's disease.
Time Frame: 19 months and 7 days
Measure: Count of Participants; unit: Participants
Arm/Group | HPV-16 E6 mTCR PBL 1x10^9 + HD IL-2 | HPV-16 E6 mTCR PBL 1x10^10 + HD IL-2 | HPV-16 E6 mTCR PBL 1x10^11 + HD IL-2 | HPV-16 E6 mTCR PBL >1x10^11 up to 2x10^11 + HD IL-2 | HPV-16 E6 mTCR PBL MTD + HD IL-2
Number analyzed (Participants) | 1 | 2 | 1 | 6 | 2
Participants | 0 | 0 | 0 | 0 | 0

6. Secondary Outcome: Percentage of Cluster of Differentiation 3 (CD3+) Cells That Are E6 T-Cell Receptor Memory of Circulating T-Cells in Responders and Non-responders
Description: Detection of E6 TCR T cells in patients peripheral blood leukocytes (PBL)/apheresis samples by flow cytometry.
Time Frame: One month after treatment
Population: One patient in group HPV-16 E6 mTCR PBL 1x10^10 + HD IL-2 did not have research blood collected at one month post infusion, and thus could not examine the cells for that patient at that time point.
Measure: Mean (95% Confidence Interval); unit: percentage of cells
Arm/Group | HPV-16 E6 mTCR PBL 1x10^9 + HD IL-2 | HPV-16 E6 mTCR PBL 1x10^10 + HD IL-2 | HPV-16 E6 mTCR PBL 1x10^11 + HD IL-2 | HPV-16 E6 mTCR PBL >1x10^11 up to 2x10^11 + HD IL-2 | HPV-16 E6 mTCR PBL MTD + HD IL-2
Number analyzed (Participants) | 1 | 1 | 1 | 6 | 2
percentage of cells
  Responders | NA — There were no responders in this group so that means they did not have a mean percentage of E6 TCR cells at one month. | NA — There were no responders in this group so that means they did not have a mean percentage of E6 TCR cells at one month. | NA — There were no responders in this group so that means they did not have a mean percentage of E6 TCR cells at one month. | 38 [30.1 to 45.9] | NA [NA to NA] — There were no responders in this group so that means they did not have a mean percentage of E6 TCR cells at one month.
  Non-responders | 30.7 [30.7 to 30.7] | 4.4 [4.4 to 4.4] | 12.6 [12.6 to 12.6] | 29.9 [10.4 to 44.4] | 37.1 [21.7 to 52.5]

7. Secondary Outcome: Expression of Programmed Cell Death 1 (PD-1) by Circulating E6 T-Cell Receptor (TCR) T-Cells
Description: Presence of PD-1 on circulating lymphocytes by flow cytometry one month after treatment.
Time Frame: one month after treatment
Population: as for outcome 6
Measure: Mean (Full Range); unit: % PD-1 circulating lymphocytes
Arm/Group | HPV-16 E6 mTCR PBL 1x10^9 + HD IL-2 | HPV-16 E6 mTCR PBL 1x10^10 + HD IL-2 | HPV-16 E6 mTCR PBL 1x10^11 + HD IL-2 | HPV-16 E6 mTCR PBL >1x10^11 up to 2x10^11 + HD IL-2 | HPV-16 E6 mTCR PBL MTD + HD IL-2
Number analyzed (Participants) | 1 | 1 | 1 | 6 | 2
% PD-1 circulating lymphocytes | 1 [1 to 1] | 2 [2 to 2] | 3 [3 to 3] | 1 [0 to 3.6] | 2.2 [0.5 to 3.9]

ADVERSE EVENTS:
Time Frame: 19 months and 7 days
Groups:
- HPV-16 E6 mTCR PBL MTD + HD IL-2-Retreatment: patients will receive cyclophosphamide and fludarabine followed by infusion of the human papilloma virus (HPV) E6 T cell receptor (TCR), followed by high dose aldesleukin
  Fludarabine: Patients will receive Fludarabine 25 mg/m^2/day for 5 days.
  Cyclophosphamide: Patients will receive Cyclophosphamide 60 mg/kg/day x 2 days
  E6 TCR: On day 0, cells will be infused intravenously (IV) over 20-30 minute (between 1 and 4 days after the last dose of fludarabine)
  Aldesleukin: Aldesleukin 720,000 IU/kg IV (based on total body weight) over 15 minutes approximately every 8 hours beginning within 24 hours of cell infusion and continuing for up to 5 days (maximum of 15 doses).
Arm/Group | HPV-16 E6 mTCR PBL 1x10^9 + HD IL-2 | HPV-16 E6 mTCR PBL 1x10^10 + HD IL-2 | HPV-16 E6 mTCR PBL 1x10^11 + HD IL-2 | HPV-16 E6 mTCR PBL >1x10^11 up to 2x10^11 + HD IL-2 | HPV-16 E6 mTCR PBL MTD + HD IL-2 | HPV-16 E6 mTCR PBL MTD + HD IL-2-Retreatment
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/2 | 0/1 | 0/6 | 0/2 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1 | 1/2 | 0/1 | 2/6 | 2/2 | 0/1
Other Adverse Events (participants affected / at risk) | 1/1 | 2/2 | 1/1 | 6/6 | 2/2 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HPV-16 E6 mTCR PBL 1x10^9 + HD IL-2 (N=1) | HPV-16 E6 mTCR PBL 1x10^10 + HD IL-2 (N=2) | HPV-16 E6 mTCR PBL 1x10^11 + HD IL-2 (N=1) | HPV-16 E6 mTCR PBL >1x10^11 up to 2x10^11 + HD IL-2 (N=6) | HPV-16 E6 mTCR PBL MTD + HD IL-2 (N=2) | HPV-16 E6 mTCR PBL MTD + HD IL-2-Retreatment (N=1)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hemorrhage, pulmonary/upper respiratory::Bronchopulmonary NOS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Obstruction/stenosis of airway::Bronchus (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Prolonged intubation after pulmonary resection (>24 hrs after surgery) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infection (documented clinically or microbiologically) (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) — with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L)::Blood
Febrile neutropenia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) — (fever of unknown origin without clinically or microbiologically documented infection)(ANC <1.0 x 10e9/L, fever >=38.5 degrees C)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HPV-16 E6 mTCR PBL 1x10^9 + HD IL-2 (N=1) | HPV-16 E6 mTCR PBL 1x10^10 + HD IL-2 (N=2) | HPV-16 E6 mTCR PBL 1x10^11 + HD IL-2 (N=1) | HPV-16 E6 mTCR PBL >1x10^11 up to 2x10^11 + HD IL-2 (N=6) | HPV-16 E6 mTCR PBL MTD + HD IL-2 (N=2) | HPV-16 E6 mTCR PBL MTD + HD IL-2-Retreatment (N=1)
Fatigue (General disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hemoglobin (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 1 (1) | 4 (4) | 2 (2) | 1 (1)
Infection (documented clinically and microbiologically) (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — with Grade 3 or 4 neutrophils (ANC<1.0x10e9/L)::Blood
Lymphopenia (Blood and lymphatic system disorders) | 1 (1) | 2 (2) | 1 (1) | 6 (6) | 2 (2) | 1 (1)
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 1 (1) | 2 (2) | 1 (1) | 6 (6) | 2 (2) | 1 (1)
Platelets (Blood and lymphatic system disorders) | 1 (1) | 2 (2) | 1 (1) | 6 (6) | 2 (2) | 1 (1)
Bilirubin (hyperbilirubinemia) (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Febrile neutropenia (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 0 (0) — (fever of unknown origin without clinically or microbiologically documented infection)(ANC<1.0 x 10e9/L, fever>=38.5 degrees C)
Psychosis (hallucinations/delusions) (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Creatinine (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Supraventricular and nodal arrhythmia::Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Syncope (fainting) (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal/Genitourinary - Other, Acute renal injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No